CLINICAL TRIAL: NCT02760498
Title: A Phase 2 Study of REGN2810, a Fully Human Monoclonal Antibody to Programmed Death-1 (PD-1), in Patients With Advanced Cutaneous Squamous Cell Carcinoma
Brief Title: Study of REGN2810 in Patients With Advanced Cutaneous Squamous Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R2810-ONC-1540; 2016-000105-36 (EudraCT Number)
Record Dates: First submitted 2016-04-08; First posted 2016-05-03 (Estimated); Results first posted 2024-12-11 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Advanced Cutaneous Squamous Cell Carcinoma
Keywords: Metastatic CSCC; Unresectable locally advanced CSCC
MeSH Terms: interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Group 1 (Participants With mCSCC): Cemiplimab 3 mg/kg Q2W (Experimental): Participants received cemiplimab 3 milligrams (mg)/kilogram (kg) intravenously (IV) every 2 weeks (Q2W) during each 8-week treatment cycle, for up to 96 weeks (12 cycles).
  Interventions: Drug: cemiplimab
- Group 2 (Participants With laCSCC): Cemiplimab 3 mg/kg Q2W (Experimental): Participants received cemiplimab 3 mg/kg IV Q2W during each 8-week treatment cycle, for up to 96 weeks (12 cycles).
  Interventions: Drug: cemiplimab
- Group 3 (Participants With mCSCC): Cemiplimab 350 mg Q3W (Experimental): Participants received cemiplimab 350 mg IV every 3 weeks (Q3W) during each 9-week treatment cycle, for up to 54 weeks (6 cycles).
  Interventions: Drug: cemiplimab
- Group 4 (Participants With mCSCC and laCSCC): Cemiplimab 600 mg Q4W (Experimental): Participants received cemiplimab 600 mg IV every 4 weeks (Q4W) during each 8-week treatment cycle, for up to 48 weeks (6 cycles).
  Interventions: Drug: cemiplimab
- Group 5 (Participants With mCSCC and laCSCC): Cemiplimab SC + 350 mg Q3W (Experimental): Participants received a single subcutaneous (SC) dose of cemiplimab followed by cemiplimab 350 mg IV Q3W during each 9-week treatment cycle, for up to 54 weeks (6 cycles).
  Interventions: Drug: cemiplimab
- Group 6 (Participants With mCSCC and laCSCC): Cemiplimab 350 mg Q3W (Experimental): Participants received cemiplimab 350 mg IV Q3W during each 9-week treatment cycle, for up to 108 weeks (12 cycles).
  Interventions: Drug: cemiplimab

INTERVENTIONS:
Drug: cemiplimab
  Other Names: REGN2810; Libtayo

SUMMARY:
The goals of this study are to evaluate the clinical benefit and safety of cemiplimab in participants with metastatic (nodal or distant) Cutaneous Squamous Cell Carcinoma (CSCC), or unresectable locally advanced CSCC.

ELIGIBILITY:
Key Inclusion Criteria:

* At least 1 measurable lesion
* Eastern Cooperative Oncology Group (ECOG) performance status ≤1
* Adequate bone marrow function
* Adequate renal function
* Adequate hepatic function
* Archived or newly obtained tumor material
* Patients must consent to undergo biopsies of CSCC lesions (Groups 2, 4, and 6)
* Surgical or radiological treatment of lesions contraindicated

Key Exclusion Criteria:

* Ongoing or recent (within 5 years) evidence of significant autoimmune disease that required treatment with systemic immunosuppressive treatments, which may suggest risk for immune-related adverse events
* Prior treatment with an agent that blocks the PD-1/PD-L1pathway
* Prior treatment with a BRAF inhibitor
* Prior treatment with other immune-modulating agents within fewer than 4 weeks prior to the first dose of cemiplimab, or associated with immune-mediated adverse events that were ≥ grade 1 within 90 days prior to the first dose of cemiplimab, or associated with toxicity that resulted in discontinuation of the immune-modulating agent. Examples of immune-modulating agents include therapeutic vaccines, cytokine treatments, or agents that target cytotoxic T-lymphocyte antigen 4 (CTLA-4), 4-1BB (CD137), or OX-40.
* Untreated brain metastasis(es) that may be considered active
* Immunosuppressive corticosteroid doses (>10 mg prednisone daily or equivalent) within 4 weeks prior to the first dose of cemiplimab
* Infection with human immunodeficiency virus (HIV) and/or chronic/active infection with hepatitis B virus or hepatitis C virus
* History of non-infectious pneumonitis within the last 5 years
* Allergic reactions or acute hypersensitivity reaction attributed to antibody treatments
* Known allergy to doxycycline or tetracycline
* Patients with a history of solid organ transplant
* Any medical co-morbidity, physical examination finding, or metabolic dysfunction, or clinical laboratory abnormality that renders the patient unsuitable

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Actual)
Dates: Start 2016-04-07 (Actual); Primary Completion 2023-10-18 (Actual); Study Completion 2023-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (78):
- United States (26):
  - University of Arizona Cancer Center, Phoenix, Arizona
  - Mayo Clinic, Phoenix, Arizona
  - City of Hope Hospital, Duarte, California
  - University of California, Los Angeles, Los Angeles, California
  - Stanford University, Redwood City, California
  - University of California, San Diego, San Diego, California
  - University of Colorado, Denver, Aurora, Colorado
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - Norton Cancer Institute, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - St. Louis University, St Louis, Missouri
  - Washington University in St. Louis, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - New York University, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Cleveland Clinic, Cleveland, Ohio
  - St. Luke's Hematology Oncology Specialists, Easton, Pennsylvania
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Dermatology and Laser Center of Charleston, Charleston, South Carolina
  - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
- Australia (10):
  - The Canberra Hospital, Garran, Australian Capital Territory
  - Gosford Hospital, Gosford, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Royal Brisbane & Women's Hospital, Herston, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Adelaide Cancer Centre, Kurralta Park, South Australia
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Border Medical Oncology, Wodonga, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Brazil (6):
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Liga Paranaense de Combate Ao Cancer - Hospital Erasto Gaertner, Curitiba
  - Fundação São Francisco Xavier-Hospital Márcio Cunha, Ipatinga
  - Animi, Lages
  - Fundação Antônio Prudente - AC Camargo Câncer Center, São Paulo
  - Instituto do Cancer do Estado de São Paulo ICESP, São Paulo
- France (11):
  - Hôpital Claude Huriez, Lille, Nord
  - Hopital Avicenne, Bobigny
  - Hôpital Saint-André, Bordeaux
  - CHU Dijon Bourgogne, Dijon
  - CHRU Grenoble, Grenoble
  - Hopitaux de La Timone, Marseille
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - Hopital Cochin, Paris
  - Hôpital Saint Louis, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Institut Gustave Roussy, Villejuif
- Germany (8):
  - Universitätsklinikum Tübingen, Tübingen, Baden-Wurttemberg
  - LMU Klinikum der Universität München, Munich, Bavaria
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Universitätsklinikum Carl Gustav Carus, Dresden, Saxony
  - Universitatsklinikum Schleswig-Holstein, Kiel, Schleswig-Holstein
  - Charitè Campus Mitte, Berlin
  - SRH Wald-Klinikum Gera, Gera
- Andreas Sygros Hosptial-University of Athen, Athens, Greece
- Italy (6):
  - Istituto Nazionale Per Lo Studio E La Cura Dei Tumori Fondazione Giovanni Pascale, Napoli, Campania
  - Istituto Oncologico Veneto - I.R.C.C.S., Padua, Veneto
  - ASST degli Spedali Civili di Brescia - Spedali Civili di Brescia, Brescia
  - Ospedale San Salvatore, L’Aquila
  - Istituto Europeo Di Oncologia, Milan
  - Fondazione Policlinico Universitario A Gemelli, Roma
- Spain (10):
  - ICO l'Hospitalet - Hospital Duran i Reynals, L'Hospitalet de Llobregat, Barelona
  - Hospital Clinic de Barcelona, Barcelona, Catalonia
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario Germans Trias i Pujol, Barcelona
  - C.H. Regional Reina Sofia - PPDS, Córdoba
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Marques de Valdecilla, Santander
  - Fundacion Instituto Valenciano de Oncología, Valencia

REFERENCES:
- [Derived] Rischin D, Hughes BGM, Basset-Seguin N, Schadendorf D, Bowyer S, Trabelsi Messai S, Meier F, Eigentler TK, Casado Echarren V, Stein B, Beylot-Barry M, Dalac S, Dreno B, Migden MR, Hauschild A, Schmults CD, Lim AM, Yoo SY, Paccaly AJ, Papachristos A, Nguyen JH, Okoye E, Seebach F, Booth J, Lowy I, Fury MG, Guminski A. High response rate with extended dosing of cemiplimab in advanced cutaneous squamous cell carcinoma. J Immunother Cancer. 2024 Mar 11;12(3):e008325. doi: 10.1136/jitc-2023-008325. PMID 38471711
- [Derived] Rischin D, Khushalani NI, Schmults CD, Guminski A, Chang ALS, Lewis KD, Lim AM, Hernandez-Aya L, Hughes BGM, Schadendorf D, Hauschild A, Thai AA, Stankevich E, Booth J, Yoo SY, Li S, Chen Z, Okoye E, Chen CI, Mastey V, Sasane M, Lowy I, Fury MG, Migden MR. Integrated analysis of a phase 2 study of cemiplimab in advanced cutaneous squamous cell carcinoma: extended follow-up of outcomes and quality of life analysis. J Immunother Cancer. 2021 Aug;9(8):e002757. doi: 10.1136/jitc-2021-002757. PMID 34413166
- [Derived] Paccaly AJ, Migden MR, Papadopoulos KP, Yang F, Davis JD, Rippley RK, Lowy I, Fury MG, Stankevich E, Rischin D. Fixed Dose of Cemiplimab in Patients with Advanced Malignancies Based on Population Pharmacokinetic Analysis. Adv Ther. 2021 May;38(5):2365-2378. doi: 10.1007/s12325-021-01638-5. Epub 2021 Mar 25. PMID 33768419
- [Derived] Rischin D, Migden MR, Lim AM, Schmults CD, Khushalani NI, Hughes BGM, Schadendorf D, Dunn LA, Hernandez-Aya L, Chang ALS, Modi B, Hauschild A, Ulrich C, Eigentler T, Stein B, Pavlick AC, Geiger JL, Gutzmer R, Alam M, Okoye E, Mathias M, Jankovic V, Stankevich E, Booth J, Li S, Lowy I, Fury MG, Guminski A. Phase 2 study of cemiplimab in patients with metastatic cutaneous squamous cell carcinoma: primary analysis of fixed-dosing, long-term outcome of weight-based dosing. J Immunother Cancer. 2020 Jun;8(1):e000775. doi: 10.1136/jitc-2020-000775. PMID 32554615
- [Derived] Migden MR, Khushalani NI, Chang ALS, Lewis KD, Schmults CD, Hernandez-Aya L, Meier F, Schadendorf D, Guminski A, Hauschild A, Wong DJ, Daniels GA, Berking C, Jankovic V, Stankevich E, Booth J, Li S, Weinreich DM, Yancopoulos GD, Lowy I, Fury MG, Rischin D. Cemiplimab in locally advanced cutaneous squamous cell carcinoma: results from an open-label, phase 2, single-arm trial. Lancet Oncol. 2020 Feb;21(2):294-305. doi: 10.1016/S1470-2045(19)30728-4. Epub 2020 Jan 14. PMID 31952975
- [Derived] Migden MR, Rischin D, Schmults CD, Guminski A, Hauschild A, Lewis KD, Chung CH, Hernandez-Aya L, Lim AM, Chang ALS, Rabinowits G, Thai AA, Dunn LA, Hughes BGM, Khushalani NI, Modi B, Schadendorf D, Gao B, Seebach F, Li S, Li J, Mathias M, Booth J, Mohan K, Stankevich E, Babiker HM, Brana I, Gil-Martin M, Homsi J, Johnson ML, Moreno V, Niu J, Owonikoko TK, Papadopoulos KP, Yancopoulos GD, Lowy I, Fury MG. PD-1 Blockade with Cemiplimab in Advanced Cutaneous Squamous-Cell Carcinoma. N Engl J Med. 2018 Jul 26;379(4):341-351. doi: 10.1056/NEJMoa1805131. Epub 2018 Jun 4. PMID 29863979
- See also: A Plain Language Summary is available on TrialSummaries.com — https://www.trialsummaries.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 432 participants with advanced cutaneous squamous cell carcinoma (CSCC) (metastatic CSCC [mCSCC] or locally advanced CSCC [laCSCC]) were enrolled.
Groups:
- Group 1 (Participants With mCSCC): Cemiplimab 3 mg/kg IV Q2W: Participants received cemiplimab 3 milligrams (mg)/kilogram (kg) intravenously (IV) every 2 weeks (Q2W) during each 8-week treatment cycle, for up to 96 weeks (12 cycles).
- Group 2 (Participants With laCSCC): Cemiplimab 3 mg/kg IV Q2W: Participants received cemiplimab 3 mg/kg IV Q2W during each 8-week treatment cycle, for up to 96 weeks (12 cycles).
- Group 3 (Participants With mCSCC): Cemiplimab 350 mg IV Q3W: Participants received cemiplimab 350 mg IV every 3 weeks (Q3W) during each 9-week treatment cycle, for up to 54 weeks (6 cycles).
- Group 4 (Participants With mCSCC and laCSCC): Cemiplimab 600 mg IV Q4W: Participants received cemiplimab 600 mg IV every 4 weeks (Q4W) during each 8-week treatment cycle, for up to 48 weeks (6 cycles).
- Group 5 (Participants With mCSCC and laCSCC): Cemiplimab 438 mg SC + 350 mg IV Q3W: Participants received a single 438 mg subcutaneous (SC) dose of cemiplimab followed by cemiplimab 350 mg IV Q3W during each 9-week treatment cycle, for up to 54 weeks (6 cycles).
- Group 6 (Participants With mCSCC and laCSCC): Cemiplimab 350 mg IV Q3W: Participants received cemiplimab 350 mg IV Q3W during each 9-week treatment cycle, for up to 108 weeks (12 cycles).
Period: Overall Study
Arm/Group | Group 1 (Participants With mCSCC): Cemiplimab 3 mg/kg IV Q2W | Group 2 (Participants With laCSCC): Cemiplimab 3 mg/kg IV Q2W | Group 3 (Participants With mCSCC): Cemiplimab 350 mg IV Q3W | Group 4 (Participants With mCSCC and laCSCC): Cemiplimab 600 mg IV Q4W | Group 5 (Participants With mCSCC and laCSCC): Cemiplimab 438 mg SC + 350 mg IV Q3W | Group 6 (Participants With mCSCC and laCSCC): Cemiplimab 350 mg IV Q3W
Started | 59 | 78 | 56 | 63 | 9 | 167
Received at Least 1 Dose of Study Drug | 59 | 78 | 56 | 63 | 9 | 165
Completed Treatment | 24 | 20 | 22 | 27 | 5 | 50
Completed (Completed Study) | 19 | 28 | 22 | 24 | 3 | 64
Not Completed | 40 | 50 | 34 | 39 | 6 | 103
Not completed — Adverse Event | 3 | 3 | 1 | 1 | 0 | 6
Not completed — Death | 7 | 5 | 5 | 7 | 0 | 23
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Non-compliance with study drug | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Participant decision | 1 | 4 | 2 | 2 | 1 | 6
Not completed — Sponsor decision | 0 | 0 | 0 | 3 | 0 | 0
Not completed — Physician Decision | 3 | 4 | 1 | 4 | 0 | 2
Not completed — Disease progression | 21 | 19 | 20 | 18 | 4 | 55
Not completed — Withdrawal by Subject | 4 | 7 | 5 | 1 | 0 | 6
Not completed — Other than specified | 1 | 6 | 0 | 3 | 1 | 0
Not completed — Not treated | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) included all enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (Participants With mCSCC): Cemiplimab 3 mg/kg IV Q2W | Group 2 (Participants With laCSCC): Cemiplimab 3 mg/kg IV Q2W | Group 3 (Participants With mCSCC): Cemiplimab 350 mg IV Q3W | Group 4 (Participants With mCSCC and laCSCC): Cemiplimab 600 mg IV Q4W | Group 5 (Participants With mCSCC and laCSCC): Cemiplimab 438 mg SC + 350 mg IV Q3W | Group 6 (Participants With mCSCC and laCSCC): Cemiplimab 350 mg IV Q3W | Total
Number analyzed (Participants) | 59 | 78 | 56 | 63 | 9 | 167 | 432
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 16 | 19 | 14 | 16 | 3 | 30 | 98
  >= 65 to < 75 years | 23 | 23 | 20 | 17 | 4 | 43 | 130
  >= 75 years | 20 | 36 | 22 | 30 | 2 | 94 | 204
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 19 | 8 | 10 | 4 | 37 | 83
  Male | 54 | 59 | 48 | 53 | 5 | 130 | 349
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 1 | 1 | 0 | 4 | 9
  Not Hispanic or Latino | 58 | 75 | 55 | 62 | 8 | 147 | 405
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1 | 16 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 2 | 2 | 1 | 0 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 0 | 0 | 1
  White | 58 | 75 | 54 | 61 | 8 | 164 | 420
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) by Independent Central Review
Description: ORR was defined as percentage of participants with best overall response (BOR) of complete response (CR) or partial response (PR). For participants with metastatic disease, Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 was used to determine BOR. For participants with unresectable locally advanced disease, clinical response criteria were used. RECIST v1.1 Criteria: -CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeter (mm) <1 (centimeter (cm). -PR: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Clinical Response Criteria: -CR: All target and nontarget lesion(s) no longer visible, maintained for at least 4 weeks and no new lesions. -PR: Decrease of at least 50% in the sum the products of perpendicular longest dimensions of target lesion(s), maintained for at least 4 weeks and no new lesions.
Time Frame: Up to 108 weeks
Population: The Full Analysis Set (FAS) included all enrolled participants. Only Groups 1, 2, 3, 4, and 6 were planned for this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 (Participants With mCSCC): Cemiplimab 3 mg/kg IV Q2W | Group 2 (Participants With laCSCC): Cemiplimab 3 mg/kg IV Q2W | Group 3 (Participants With mCSCC): Cemiplimab 350 mg IV Q3W | Group 4 (Participants With mCSCC and laCSCC): Cemiplimab 600 mg IV Q4W | Group 6 (Participants With mCSCC and laCSCC): Cemiplimab 350 mg IV Q3W
Number analyzed (Participants) | 59 | 78 | 56 | 63 | 167
percentage of participants | 50.8 [37.5 to 64.1] | 44.9 [33.6 to 56.6] | 46.4 [33.0 to 60.3] | 61.9 [48.8 to 73.9] | 47.3 [39.5 to 55.2]

2. Secondary Outcome: ORR by Investigator Assessment
Description: ORR was defined as percentage of participants with BOR of CR or PR. For participants with metastatic disease, RECIST v1.1 was used to determine BOR. For participants with unresectable locally advanced disease, clinical response criteria were used. RECIST v1.1 Criteria: -CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm <1 cm. -PR: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Clinical Response Criteria: -CR: All target and nontarget lesion(s) no longer visible, maintained for at least 4 weeks and no new lesions. -PR: Decrease of at least 50% in the sum the products of perpendicular longest dimensions of target lesion(s), maintained for at least 4 weeks and no new lesions.
Time Frame: Up to 108 weeks
Population: The FAS included all enrolled participants. Only Groups 1, 2, 3, 4, and 6 were planned for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 (Participants With mCSCC): Cemiplimab 3 mg/kg IV Q2W | Group 2 (Participants With laCSCC): Cemiplimab 3 mg/kg IV Q2W | Group 3 (Participants With mCSCC): Cemiplimab 350 mg IV Q3W | Group 4 (Participants With mCSCC and laCSCC): Cemiplimab 600 mg IV Q4W | Group 6 (Participants With mCSCC and laCSCC): Cemiplimab 350 mg IV Q3W
Number analyzed (Participants) | 59 | 78 | 56 | 63 | 167
percentage of participants | 50.8 [37.5 to 64.1] | 56.4 [44.7 to 67.6] | 55.4 [41.5 to 68.7] | 63.5 [50.4 to 75.3] | 52.7 [44.8 to 60.5]

3. Secondary Outcome: Duration of Response (DOR) by Independent Central Review
Description: DOR was measured from the time measurement criteria were first met for CR/PR, whichever was recorded first, until the first date of recurrent or Progressive Disease (PD) or death due to any cause in participants with BOR of CR or PR. For participants with metastatic disease, RECIST v1.1 was used to determine BOR. For participants with unresectable locally advanced disease, clinical response criteria were used. RECIST v1.1 Criteria: -PD: At least a 20% increase in the sum of the diameters of target lesions with the sum demonstrating an absolute increase of at least 5 mm (0.5 cm), or the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Clinical Response Criteria: -PD: increase of ≥ 25% (WHO criteria) in the sum of the products of perpendicular longest dimensions of target lesion(s) and/or the appearance of new lesions.
Time Frame: Up to approximately 65 months (treatment period + follow-up including survival follow-up)
Population: The FAS included all enrolled participants. Here, 'Overall number of participants analyzed' signifies participants with confirmed CR or PR who were evaluable for this outcome measure. Only Groups 1, 2, 3, 4, and 6 were planned for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group 1 (Participants With mCSCC): Cemiplimab 3 mg/kg IV Q2W | Group 2 (Participants With laCSCC): Cemiplimab 3 mg/kg IV Q2W | Group 3 (Participants With mCSCC): Cemiplimab 350 mg IV Q3W | Group 4 (Participants With mCSCC and laCSCC): Cemiplimab 600 mg IV Q4W | Group 6 (Participants With mCSCC and laCSCC): Cemiplimab 350 mg IV Q3W
Number analyzed (Participants) | 30 | 35 | 26 | 39 | 79
months | NA [20.7 to NA] — Not reached due to insufficient number of events | 41.9 [20.5 to 54.6] | 41.3 [40.8 to 46.3] | NA [30.5 to NA] — Not reached due to insufficient number of events | 31.6 [29.5 to NA] — Not reached due to insufficient number of events

4. Secondary Outcome: DOR by Investigator Assessment
Description: DOR was measured from the time measurement criteria were first met for CR/PR, as defined in Outcome Measure 1, whichever was recorded first, until the first date of recurrent or Progressive Disease (PD) or death due to any cause in participants with BOR of CR or PR. For participants with metastatic disease, RECIST v1.1 was used to determine BOR. For participants with unresectable locally advanced disease, clinical response criteria were used. RECIST v1.1 Criteria: -PD: At least a 20% increase in the sum of the diameters of target lesions with the sum demonstrating an absolute increase of at least 5 mm (0.5 cm), or the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Clinical Response Criteria: -PD: increase of ≥ 25% (World Health Organization (WHO) criteria) in the sum of the products of perpendicular longest dimensions of target lesion(s) and/or the appearance of new lesions.
Time Frame: Up to approximately 65 months (treatment period + follow-up including survival follow-up)
Population: The FAS included all enrolled participants. Here, 'Overall number of participants analyzed' signifies participants with confirmed CR or PR that are evaluable for this outcome measure. Only Groups 1, 2, 3, 4, and 6 were planned for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group 1 (Participants With mCSCC): Cemiplimab 3 mg/kg IV Q2W | Group 2 (Participants With laCSCC): Cemiplimab 3 mg/kg IV Q2W | Group 3 (Participants With mCSCC): Cemiplimab 350 mg IV Q3W | Group 4 (Participants With mCSCC and laCSCC): Cemiplimab 600 mg IV Q4W | Group 6 (Participants With mCSCC and laCSCC): Cemiplimab 350 mg IV Q3W
Number analyzed (Participants) | 30 | 44 | 31 | 40 | 88
months | NA [30.7 to NA] — Not reached due to insufficient number of events | 41.9 [NA to NA] — Not reached due to insufficient number of events | 44.2 [25.4 to 44.2] | NA [27.1 to NA] — Not reached due to insufficient number of events | NA [29.5 to NA] — Not reached due to insufficient number of events

5. Secondary Outcome: Progression-Free Survival (PFS) by Independent Central Review
Description: PFS was measured from start of treatment until the first date of recurrent or PD, or death due to any cause. For participants with metastatic disease, RECIST v1.1 was used to determine PD. For participants with unresectable locally advanced disease, clinical response criteria were used. RECIST v1.1 Criteria: -PD: At least a 20% increase in the sum of the diameters of target lesions with the sum demonstrating an absolute increase of at least 5 mm (0.5 cm), or the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Clinical Response Criteria: -PD: increase of ≥ 25% (WHO criteria) in the sum of the products of perpendicular longest dimensions of target lesion(s) and/or the appearance of new lesions.
Time Frame: Up to approximately 65 months (treatment period + follow-up including survival follow-up)
Population: The FAS included all enrolled participants. Here, 'Overall number of participants analyzed' signifies participants who received at least one dose of cemiplimab and were evaluable for this outcome measure. Only Groups 1, 2, 3, 4, and 6 were planned for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group 1 (Participants With mCSCC): Cemiplimab 3 mg/kg IV Q2W | Group 2 (Participants With laCSCC): Cemiplimab 3 mg/kg IV Q2W | Group 3 (Participants With mCSCC): Cemiplimab 350 mg IV Q3W | Group 4 (Participants With mCSCC and laCSCC): Cemiplimab 600 mg IV Q4W | Group 6 (Participants With mCSCC and laCSCC): Cemiplimab 350 mg IV Q3W
Number analyzed (Participants) | 59 | 78 | 56 | 63 | 165
months | 18.4 [7.3 to 53.2] | 18.5 [11.1 to 43.8] | 21.7 [3.8 to 43.3] | 32.2 [16.6 to NA] — Not reached due to insufficient number of events | 16.6 [12.4 to 31.5]

6. Secondary Outcome: PFS by Investigator Assessment
Description: as for outcome 5
Time Frame: Up to approximately 65 months (treatment period + follow-up including survival follow-up)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group 1 (Participants With mCSCC): Cemiplimab 3 mg/kg IV Q2W | Group 2 (Participants With laCSCC): Cemiplimab 3 mg/kg IV Q2W | Group 3 (Participants With mCSCC): Cemiplimab 350 mg IV Q3W | Group 4 (Participants With mCSCC and laCSCC): Cemiplimab 600 mg IV Q4W | Group 6 (Participants With mCSCC and laCSCC): Cemiplimab 350 mg IV Q3W
Number analyzed (Participants) | 59 | 78 | 56 | 63 | 165
months | 16.6 [7.3 to NA] — Not reached due to insufficient number of events | 32.5 [17.1 to 43.8] | 15.2 [4.1 to 43.0] | 25.3 [8.2 to NA] — Not reached due to insufficient number of events | 16.5 [10.3 to 31.3]

7. Secondary Outcome: Overall Survival (OS)
Description: OS was measured from start of treatment until death due to any cause.
Time Frame: Up to approximately 65 months (treatment period + follow-up including survival follow-up)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group 1 (Participants With mCSCC): Cemiplimab 3 mg/kg IV Q2W | Group 2 (Participants With laCSCC): Cemiplimab 3 mg/kg IV Q2W | Group 3 (Participants With mCSCC): Cemiplimab 350 mg IV Q3W | Group 4 (Participants With mCSCC and laCSCC): Cemiplimab 600 mg IV Q4W | Group 6 (Participants With mCSCC and laCSCC): Cemiplimab 350 mg IV Q3W
Number analyzed (Participants) | 59 | 78 | 56 | 63 | 165
months | 57.7 [29.3 to NA] — Not reached due to insufficient number of events | NA [58.3 to NA] — Not reached due to insufficient number of events | 48.4 [29.5 to NA] — Not reached due to insufficient number of events | NA [28.6 to NA] — Not reached due to insufficient number of events | NA [NA to NA] — Not reached due to insufficient number of events

8. Secondary Outcome: Complete Response (CR) Rate by Independent Central Review
Description: CR rate was defined as percentage of participants with BOR of CR. For participants with metastatic disease, RECIST v1.1 was used to determine BOR. For participants with unresectable locally advanced disease, clinical response criteria were used. RECIST v1.1 Criteria: -CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm <1 cm. Clinical Response Criteria: -CR: All target and nontarget lesion(s) no longer visible, maintained for at least 4 weeks and no new lesions.
Time Frame: Up to 108 weeks
Population: The FAS included all enrolled participants. Only Groups 1, 2, 3, 4, and 6 were planned for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 (Participants With mCSCC): Cemiplimab 3 mg/kg IV Q2W | Group 2 (Participants With laCSCC): Cemiplimab 3 mg/kg IV Q2W | Group 3 (Participants With mCSCC): Cemiplimab 350 mg IV Q3W | Group 4 (Participants With mCSCC and laCSCC): Cemiplimab 600 mg IV Q4W | Group 6 (Participants With mCSCC and laCSCC): Cemiplimab 350 mg IV Q3W
Number analyzed (Participants) | 59 | 78 | 56 | 63 | 167
percentage of participants | 20.3 [11.0 to 32.8] | 12.8 [6.3 to 22.3] | 19.6 [10.2 to 32.4] | 22.2 [12.7 to 34.5] | 10.8 [6.5 to 16.5]

9. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) Global Health Status (GHS) Score
Description: EORTC QLQ-C30 is a 30-question tool used to assess the overall quality of life (QoL) in cancer participants. Items contributing to the GHS/QoL, were scored 1 ("very poor") to 7 ("excellent"). A linear transformation was applied to the raw scores so that transformed score lies between 0 to 100. A higher score indicates better global health status/functioning and a negative change from baseline indicated less improvement.
Time Frame: Baseline, Up to Cycle 12 Day 1 (Week 89)
Population: The FAS included all enrolled participants. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure and "Number Analyzed" is the number evaluable at each time point. Only Groups 1, 2, 3, and 4 were planned for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 (Participants With mCSCC): Cemiplimab 3 mg/kg IV Q2W | Group 2 (Participants With laCSCC): Cemiplimab 3 mg/kg IV Q2W | Group 3 (Participants With mCSCC): Cemiplimab 350 mg IV Q3W | Group 4 (Participants With mCSCC and laCSCC): Cemiplimab 600 mg IV Q4W
Number analyzed (Participants) | 44 | 68 | 38 | 54
score on a scale
  Cycle 2 Day 1 (C2D1): number analyzed (Participants) | 42 | 60 | 34 | 52
  Cycle 2 Day 1 (C2D1) | 0.00 (21.464) | 5.56 (18.895) | 6.86 (19.621) | 0.96 (17.670)
  C3D1: number analyzed (Participants) | 37 | 55 | 30 | 43
  C3D1 | 11.26 (19.267) | 5.30 (21.717) | 15.28 (20.655) | 3.88 (15.680)
  C4D1: number analyzed (Participants) | 36 | 39 | 29 | 38
  C4D1 | 6.25 (25.069) | 8.76 (19.585) | 13.51 (22.539) | 4.39 (15.099)
  C5D1: number analyzed (Participants) | 36 | 41 | 27 | 36
  C5D1 | 4.17 (22.316) | 8.33 (21.246) | 13.27 (21.466) | 5.79 (18.774)
  C6D1: number analyzed (Participants) | 31 | 44 | 26 | 33
  C6D1 | 5.11 (17.437) | 5.68 (28.118) | 12.18 (24.521) | 0.25 (21.599)
  C7D1: number analyzed (Participants) | 32 | 40 | 12 | 15
  C7D1 | 6.51 (17.676) | 9.17 (22.393) | 22.22 (23.659) | 4.44 (18.598)
  C8D1: number analyzed (Participants) | 29 | 33 | 11 | 15
  C8D1 | 4.60 (21.080) | 10.10 (21.425) | 30.30 (19.816) | 5.00 (25.158)
  C9D1: number analyzed (Participants) | 26 | 29 | 10 | 13
  C9D1 | 6.09 (18.938) | 6.61 (26.199) | 26.67 (24.470) | 7.69 (20.543)
  C10D1: number analyzed (Participants) | 27 | 23 | 9 | 10
  C10D1 | 12.04 (20.844) | 13.77 (26.064) | 28.70 (13.889) | 5.83 (22.923)
  C11D1: number analyzed (Participants) | 25 | 19 | 10 | 9
  C11D1 | 10.33 (28.186) | 11.40 (22.603) | 32.50 (14.407) | 14.81 (19.444)
  C12D1: number analyzed (Participants) | 24 | 17 | 9 | 9
  C12D1 | 8.33 (22.388) | 12.75 (24.494) | 27.78 (16.667) | 2.78 (26.021)

10. Secondary Outcome: Number of Participants With Any Treatment Emergent Adverse Event (TEAE)
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious Adverse Events (SAEs) were defined as death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed in this definition. Treatment-emergent adverse events (TEAEs) are defined as those not present at baseline or represent the exacerbation of a condition present at baseline during the on-treatment period or follow-up period. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Up to 108 weeks plus 105 days (5 half-lives)
Population: The Safety Analysis Set (SAF) included all enrolled participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Participants With mCSCC): Cemiplimab 3 mg/kg IV Q2W | Group 2 (Participants With laCSCC): Cemiplimab 3 mg/kg IV Q2W | Group 3 (Participants With mCSCC): Cemiplimab 350 mg IV Q3W | Group 4 (Participants With mCSCC and laCSCC): Cemiplimab 600 mg IV Q4W | Group 5 (Participants With mCSCC and laCSCC): Cemiplimab 438 mg SC + 350 mg IV Q3W | Group 6 (Participants With mCSCC and laCSCC): Cemiplimab 350 mg IV Q3W
Number analyzed (Participants) | 59 | 78 | 56 | 63 | 9 | 165
Participants | 59 | 78 | 55 | 63 | 9 | 163

11. Secondary Outcome: Peak Concentration (Cmax) of Cemiplimab
Time Frame: Up to approximately 43 months
Population: The Pharmacokinetic (PK) analysis set included all participants who had received cemiplimab and had at least 1 qualified (non-missing) post-baseline measurement of cemiplimab concentration in serum. Here, "Overall number of participants analyzed" is the number of participants evaluable for this outcome measure, and "Number analyzed" is the number of participants evaluable at each specified point.
Measure: Mean (Standard Deviation); unit: milligram per liter (mg/L)
Arm/Group | Group 1 (Participants With mCSCC): Cemiplimab 3 mg/kg IV Q2W | Group 2 (Participants With laCSCC): Cemiplimab 3 mg/kg IV Q2W | Group 3 (Participants With mCSCC): Cemiplimab 350 mg IV Q3W | Group 4 (Participants With mCSCC and laCSCC): Cemiplimab 600 mg IV Q4W | Group 5 (Participants With mCSCC and laCSCC): Cemiplimab 438 mg SC + 350 mg IV Q3W | Group 6 (Participants With mCSCC and laCSCC): Cemiplimab 350 mg IV Q3W
Number analyzed (Participants) | 58 | 75 | 52 | 62 | 9 | 162
milligram per liter (mg/L)
  After the First Dose | 108 (147) | 84.1 (105) | 132 (203) | 174 (50.1) | 52.9 (18.4) | 96.3 (56.2)
  At Steady State: number analyzed (Participants) | 38 | 58 | 33 | 41 | 7 | 104
  At Steady State | 151 (83.7) | 148 (76.6) | 151 (46.2) | 281 (235) | 174 (62.2) | 142 (78.3)

12. Secondary Outcome: Trough Concentration (Ctrough) of Cemiplimab
Time Frame: Up to approximately 43 months
Population: The PK analysis set included all participants who had received cemiplimab and had at least 1 qualified (non-missing) post-baseline measurement of cemiplimab concentration in serum. Here, "Overall number of participants analyzed" is the number of participants evaluable for this outcome measure, and "Number analyzed" is the number of participants evaluable at each specified point.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Group 1 (Participants With mCSCC): Cemiplimab 3 mg/kg IV Q2W | Group 2 (Participants With laCSCC): Cemiplimab 3 mg/kg IV Q2W | Group 3 (Participants With mCSCC): Cemiplimab 350 mg IV Q3W | Group 4 (Participants With mCSCC and laCSCC): Cemiplimab 600 mg IV Q4W | Group 5 (Participants With mCSCC and laCSCC): Cemiplimab 438 mg SC + 350 mg IV Q3W | Group 6 (Participants With mCSCC and laCSCC): Cemiplimab 350 mg IV Q3W
Number analyzed (Participants) | 53 | 71 | 46 | 58 | 9 | 143
mg/L
  After the First Dose: number analyzed (Participants) | 53 | 71 | 46 | 58 | 9 | 142
  After the First Dose | 21.5 (7.12) | 26.3 (14.3) | 33.6 (32.1) | 32.1 (10.4) | 34.1 (14.1) | 23.0 (10.9)
  At Steady State: number analyzed (Participants) | 38 | 58 | 34 | 44 | 7 | 106
  At Steady State | 69.9 (19.3) | 67.5 (29.8) | 62.7 (28.3) | 62.5 (24.1) | 65.9 (22.9) | 53.3 (20.1)

13. Secondary Outcome: Number of Participants With Treatment-Emergent Anti-cemiplimab Antibodies
Time Frame: Up to approximately 43 months
Population: The Anti-drug Antibody (ADA) population for cemiplimab included all treated participants who had at least 1 postdose ADA result for cemiplimab.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Participants With mCSCC): Cemiplimab 3 mg/kg IV Q2W | Group 2 (Participants With laCSCC): Cemiplimab 3 mg/kg IV Q2W | Group 3 (Participants With mCSCC): Cemiplimab 350 mg IV Q3W | Group 4 (Participants With mCSCC and laCSCC): Cemiplimab 600 mg IV Q4W | Group 5 (Participants With mCSCC and laCSCC): Cemiplimab 438 mg SC + 350 mg IV Q3W | Group 6 (Participants With mCSCC and laCSCC): Cemiplimab 350 mg IV Q3W
Number analyzed (Participants) | 50 | 66 | 41 | 50 | 8 | 133
Participants | 1 | 0 | 0 | 0 | 0 | 5

14. Secondary Outcome: ORR by Independent Central Review for Participants With Evaluable PD-L1 Assays
Description: ORR was defined as percentage of participants with BOR of CR or PR. Expression level of PD-L1 was assessed in tumor biopsy samples by immunohistochemistry (IHC). -CR: All target and nontarget lesion(s) no longer visible, maintained for at least 4 weeks and no new lesions. -PR: Decrease of at least 50% in the sum the products of perpendicular longest dimensions of target lesion(s), maintained for at least 4 weeks and no new lesions.
Time Frame: Up to 108 weeks
Population: The biomarker analysis set (BAS) included all participants in the FAS who had samples evaluable for PD-L1 assay. Here, 'Overall number of participants analyzed' is the number of participants who are evaluable for this outcome measure and "Number analyzed" is the number of participants in each row category. Only Group 6 was planned for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 6 (Participants With mCSCC and laCSCC): Cemiplimab 350 mg IV Q3W
Number analyzed (Participants) | 96
percentage of participants
  PD-L1 < 1%: number analyzed (Participants) | 37
  PD-L1 < 1% | 40.5 [24.8 to 57.9]
  PD-L1 >= 1%: number analyzed (Participants) | 59
  PD-L1 >= 1% | 49.2 [35.9 to 62.5]

15. Secondary Outcome: DOR by Independent Central Review for Participants With Evaluable PD-L1 Assays
Description: DOR was measured from the time measurement criteria are first met for CR/PR, as defined in Outcome Measure 13, whichever was recorded first, until the first date of recurrent or PD or death due to any cause in participants with BOR of CR or PR. Expression level of PD-L1 was assessed in tumor biopsy samples by IHC. -PD: increase of ≥ 25% (WHO criteria) in the sum of the products of perpendicular longest dimensions of target lesion(s) and/or the appearance of new lesions.
Time Frame: Up to approximately 65 months (treatment period + follow-up including survival follow-up)
Population: The biomarker analysis set (BAS) included all participants in the FAS who had samples evaluable for PD-L1 assay. Here, 'Overall number of participants analyzed' signifies participants with confirmed CR or PR that are evaluable for this outcome measure and "Number analyzed" is the number of participants in each row category. Only Group 6 was planned for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group 6 (Participants With mCSCC and laCSCC): Cemiplimab 350 mg IV Q3W
Number analyzed (Participants) | 44
months
  PD-L1 < 1%: number analyzed (Participants) | 15
  PD-L1 < 1% | 31.6 [12.6 to NA] — Not reached due to insufficient number of events
  PD-L1 >= 1%: number analyzed (Participants) | 29
  PD-L1 >= 1% | NA [NA to NA] — Not reached due to insufficient number of events

16. Secondary Outcome: PFS by Independent Central Review for Participants With Evaluable PD-L1 Assays
Description: PFS was measured from time of enrollment until the first date of recurrent or progressive disease, or death due to any cause. Expression level of PD-L1 was assessed in tumor biopsy samples. -PD: increase of ≥ 25% (WHO criteria) in the sum of the products of perpendicular longest dimensions of target lesion(s) and/or the appearance of new lesions.
Time Frame: Up to approximately 65 months (treatment period + follow-up including survival follow-up)
Population: The biomarker analysis set (BAS) included all participants in the FAS who had samples evaluable for PD-L1 assay. Here, 'Overall number of participants analyzed' signifies participants who are evaluable for this outcome measure and "Number analyzed" is the number of participants in each row category. Only Group 6 was planned for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group 6 (Participants With mCSCC and laCSCC): Cemiplimab 350 mg IV Q3W
Number analyzed (Participants) | 96
months
  PD-L1 < 1%: number analyzed (Participants) | 37
  PD-L1 < 1% | 10.7 [3.0 to 15.3]
  PD-L1 >= 1%: number analyzed (Participants) | 59
  PD-L1 >= 1% | 16.6 [4.0 to NA] — Not reached due to insufficient number of events

ADVERSE EVENTS:
Time Frame: From signing of informed consent through end of study up to approximately 65 months (treatment period + follow-up including survival follow-up)
Description: The Safety Analysis Set (SAF) included all enrolled participants who received any study drug.
Groups:
- Group 6a (Participants With mCSCC and laCSCC): Cemiplimab 350 mg IV Q3W to 350 mg SC Q3W: Participants in group 6 who received cemiplimab 350 mg IV Q3W and opted to switch to cemiplimab 350 mg SC Q3W for up to a total (IV + SC) of 108 weeks.
- Group 6b (Participants With mCSCC and laCSCC): Cemiplimab 350 mg IV Q3W to 1050 mg SC Q6W: Participants in group 6 who received cemiplimab 350 mg IV Q3W and opted to switch to cemiplimab 1050 mg SC Q6W for up to a total (IV + SC) of 108 weeks.
Arm/Group | Group 1 (Participants With mCSCC): Cemiplimab 3 mg/kg IV Q2W | Group 2 (Participants With laCSCC): Cemiplimab 3 mg/kg IV Q2W | Group 3 (Participants With mCSCC): Cemiplimab 350 mg IV Q3W | Group 4 (Participants With mCSCC and laCSCC): Cemiplimab 600 mg IV Q4W | Group 5 (Participants With mCSCC and laCSCC): Cemiplimab 438 mg SC + 350 mg IV Q3W | Group 6 (Participants With mCSCC and laCSCC): Cemiplimab 350 mg IV Q3W | Group 6a (Participants With mCSCC and laCSCC): Cemiplimab 350 mg IV Q3W to 350 mg SC Q3W | Group 6b (Participants With mCSCC and laCSCC): Cemiplimab 350 mg IV Q3W to 1050 mg SC Q6W
All-Cause Mortality (participants affected / at risk) | 27/59 | 19/78 | 26/56 | 23/63 | 2/9 | 59/165 | 2/12 | 0/7
Serious Adverse Events (participants affected / at risk) | 24/59 | 28/78 | 23/56 | 35/63 | 2/9 | 85/165 | 4/12 | 1/7
Other Adverse Events (participants affected / at risk) | 56/59 | 75/78 | 49/56 | 59/63 | 9/9 | 147/165 | 9/12 | 5/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (Participants With mCSCC): Cemiplimab 3 mg/kg IV Q2W (N=59) | Group 2 (Participants With laCSCC): Cemiplimab 3 mg/kg IV Q2W (N=78) | Group 3 (Participants With mCSCC): Cemiplimab 350 mg IV Q3W (N=56) | Group 4 (Participants With mCSCC and laCSCC): Cemiplimab 600 mg IV Q4W (N=63) | Group 5 (Participants With mCSCC and laCSCC): Cemiplimab 438 mg SC + 350 mg IV Q3W (N=9) | Group 6 (Participants With mCSCC and laCSCC): Cemiplimab 350 mg IV Q3W (N=165) | Group 6a (Participants With mCSCC and laCSCC): Cemiplimab 350 mg IV Q3W to 350 mg SC Q3W (N=12) | Group 6b (Participants With mCSCC and laCSCC): Cemiplimab 350 mg IV Q3W to 1050 mg SC Q6W (N=7)
Pneumonia (Infections and infestations) | 2 (2) | 5 (6) | 0 (0) | 3 (3) | 0 (0) | 7 (9) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 4 (6) | 2 (2) | 1 (1) | 1 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Encephalitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Extradural abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoas abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abscess bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected skin ulcer (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meningitis aseptic (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 4 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Follicular lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Drug withdrawal syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sudden death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carotid artery aneurysm (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Focal dyscognitive seizures (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vasogenic cerebral oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ulcerative keratitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Overflow diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza A virus test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General physical condition abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Troponin I increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arterial haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated hypophysitis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adjustment disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Autoimmune nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (Participants With mCSCC): Cemiplimab 3 mg/kg IV Q2W (N=59) | Group 2 (Participants With laCSCC): Cemiplimab 3 mg/kg IV Q2W (N=78) | Group 3 (Participants With mCSCC): Cemiplimab 350 mg IV Q3W (N=56) | Group 4 (Participants With mCSCC and laCSCC): Cemiplimab 600 mg IV Q4W (N=63) | Group 5 (Participants With mCSCC and laCSCC): Cemiplimab 438 mg SC + 350 mg IV Q3W (N=9) | Group 6 (Participants With mCSCC and laCSCC): Cemiplimab 350 mg IV Q3W (N=165) | Group 6a (Participants With mCSCC and laCSCC): Cemiplimab 350 mg IV Q3W to 350 mg SC Q3W (N=12) | Group 6b (Participants With mCSCC and laCSCC): Cemiplimab 350 mg IV Q3W to 1050 mg SC Q6W (N=7)
Diarrhoea (Gastrointestinal disorders) | 17 (29) | 23 (42) | 13 (18) | 17 (23) | 3 (3) | 39 (58) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 14 (17) | 20 (25) | 12 (12) | 6 (6) | 2 (2) | 33 (37) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 12 (12) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (8) | 11 (13) | 8 (8) | 6 (6) | 1 (1) | 17 (26) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 10 (12) | 10 (11) | 10 (11) | 15 (16) | 0 (0) | 22 (25) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 4 (4) | 3 (4) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 5 (5) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Poor dental condition (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 15 (18) | 34 (41) | 17 (19) | 14 (15) | 1 (1) | 44 (49) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 6 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 6 (8) | 0 (0) | 6 (8) | 0 (0) | 15 (16) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 4 (4) | 4 (4) | 6 (6) | 7 (7) | 0 (0) | 16 (18) | 1 (2) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 0 (0) | 26 (35) | 1 (1) | 0 (0)
Catheter site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 9 (9) | 0 (0) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Terminal agitation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (14) | 23 (29) | 7 (8) | 16 (20) | 1 (1) | 43 (55) | 1 (2) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 4 (4) | 12 (15) | 7 (7) | 8 (13) | 0 (0) | 17 (30) | 2 (2) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 11 (18) | 11 (15) | 10 (13) | 12 (17) | 3 (3) | 11 (13) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (6) | 8 (9) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9 (11) | 8 (13) | 7 (8) | 8 (10) | 4 (7) | 18 (23) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (4) | 6 (13) | 0 (0) | 10 (26) | 2 (5) | 1 (1)
Tumour pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 8 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 8 (9) | 7 (7) | 4 (4) | 7 (7) | 1 (1) | 22 (23) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 7 (9) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 7 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (5) | 7 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 6 (6) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 5 (5) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (16) | 11 (12) | 10 (13) | 11 (12) | 1 (3) | 24 (32) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (7) | 8 (8) | 6 (6) | 6 (6) | 0 (0) | 16 (17) | 2 (2) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 5 (6) | 0 (0) | 0 (0) | 1 (1) | 11 (12) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (7) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 5 (5) | 10 (10) | 0 (0) | 0 (0) | 1 (1) | 12 (15) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 4 (5) | 8 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 6 (6) | 4 (4) | 0 (0) | 1 (1) | 12 (13) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 4 (6) | 5 (5) | 5 (5) | 7 (10) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Red blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 16 (18) | 5 (5) | 7 (9) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 6 (6) | 3 (3) | 6 (7) | 1 (1) | 11 (12) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 6 (13) | 9 (12) | 5 (6) | 8 (12) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 4 (6) | 7 (7) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 6 (13) | 5 (11) | 0 (0) | 5 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 4 (7) | 4 (5) | 0 (0) | 7 (12) | 0 (0) | 10 (16) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 13 (14) | 4 (4) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 4 (6) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infected cyst (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (9) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 5 (5) | 0 (0) | 0 (0) | 5 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 7 (9) | 8 (13) | 8 (8) | 8 (13) | 1 (1) | 11 (13) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (6) | 10 (15) | 3 (5) | 6 (16) | 0 (0) | 14 (32) | 2 (6) | 2 (5)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 12 (25) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (10) | 4 (6) | 3 (3) | 0 (0) | 0 (0) | 10 (19) | 2 (2) | 0 (0)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 11 (12) | 7 (8) | 3 (4) | 7 (7) | 1 (1) | 15 (16) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 8 (9) | 5 (5) | 0 (0) | 5 (5) | 0 (0) | 13 (13) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myoclonus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 6 (6) | 9 (9) | 7 (7) | 0 (0) | 2 (2) | 14 (15) | 1 (1) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thyroid mass (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 5 (5) | 4 (4) | 4 (6) | 4 (6) | 1 (1) | 14 (16) | 2 (2) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 4 (5) | 0 (0) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radiation skin injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scar (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 8 (8) | 3 (3) | 0 (0) | 1 (1) | 9 (9) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 6 (6) | 7 (11) | 0 (0) | 0 (0) | 0 (0) | 12 (18) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otorrhoea (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the Sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2021-09-09): https://cdn.clinicaltrials.gov/large-docs/98/NCT02760498/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-12): https://cdn.clinicaltrials.gov/large-docs/98/NCT02760498/SAP_001.pdf